CLINICAL TRIAL: NCT04355572
Title: Evaluation of the Clinical and Psychological Impact of Vitamin D Replacement in Adolescent Females at Risk for Polycystic Ovarian Syndrome (PCOS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000028054; 000 (Other: CTGTY)
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Polycystic Ovarian Syndrome in Adolescent Females; Vitamin D Deficiency
Keywords: Anti-Mullerian Hormone (AMH)
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will be blinded to treatment modality until the end of the trial period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D Supplement (Experimental): Patients will take vitamin D tablet with 4,000IU daily for 6 months.
  Interventions: Drug: Vitamin D 4000IU daily
- Placebo (Placebo Comparator): Patients will take placebo for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D 4000IU daily — Randomized to receive vitamin D 4000IU daily
  Arms: Vitamin D Supplement
Drug: Placebo — Randomized to placebo daily
  Arms: Placebo

SUMMARY:
This study is a double blind, placebo controlled, randomized trial of study subjects with PCOS and low vitamin D to 2 groups- placebo and vitamin D replacement. Participants and investigators will be blinded to treatment modality until the end of the trial period

DETAILED DESCRIPTION:
Patients referred to the pediatric endocrinology clinic or adolescent gynecology clinic at Yale New Haven Children Hospital with a primary complaint of hirsutism, acne, or amenorrhea and/or oligomenorrhea persisting 2 years after their menarche will be evaluated for polycystic ovarian syndrome through history, physical exam, pelvic ultrasound, and laboratory evaluation, to include androgen testing, thyroid testing, female hormone testing, and diabetic risk testing (this is standard of care). A vitamin D level will also be drawn. While vitamin D level is not currently part of the diagnostic algorithm for PCOS, it is not unreasonable to check in patients in which there is concern for an endocrine disorder. If the patient meets Rotterdam criteria and their serum vitamin D level is between 6 and 29 ng/mL, the patient and their guardian(s) will be approached for inclusion in our study by the physician or dedicated research nursing staff.

If patient and guardian agree to participate and sign a consent / assent form, the patient will then be randomized to receive vitamin D supplement versus placebo and will be followed for 6 months on their randomized replacement with repeat laboratory testing of AMH, vitamin D, lipid profile, glucose and insulin testing, androgen testing, and female hormone testing at the randomization, 3 months and at the end of the course of the trial(6 months). Patients with vitamin D levels 5ng/mL or less will not be randomized, they will be given recommended treatment. Depressive symptoms will be assessed at time of randomization, 3 months post randomization, and 6 months post randomization using the Beck Depression Inventory-II, the gold standard self-report depression inventory. A depression screen is currently administered to all adolescents seen at Yale New Haven Children Hospital outpatient clinics with a protocol for patients who report clinically significant levels of depression. This protocol will remain in place and will not be altered during this research study.

After post-trial testing, patients will be unblinded and patients who still have vitamin D below threshold will be offered vitamin D treatment.

Aim 1: To investigate the effect of vitamin D replacement upon biochemical parameters of polycystic ovarian syndrome (PCOS) in adolescent female patients. Hypothesis: Replacement of vitamin D to normal levels in adolescents with PCOS and/or at risk for PCOS and low levels of vitamin D will lower serum androgen and anti-mullerian hormone (AMH) levels.

Aim 2: To investigate the effect of vitamin D replacement on clinical features of PCOS in adolescent female patients. Hypothesis: Replacement of vitamin D in adolescents with PCOS and/or at risk for PCOS and low levels of vitamin D will improve symptoms of menstrual irregularities, acne, and hirsutism.

Aim3: To investigate the effect of vitamin D replacement on depressive symptoms in adolescent female patients with PCOS. Hypothesis: Replacement of vitamin D in adolescents with PCOS or at risk for PCOS and low levels of serum vitamin D will improve symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

- Postmenarchal adolescent females aged 13-21 who meet modified Rotterdam criteria for PCOS, with a serum vitamin D level between 6-29 ng/mL.

Exclusion Criteria:

* Other causes for hyperandrogenism,
* Chronic renal diseases,
* Acquired or inherited calcium and vitamin D metabolic disorders.

Ages: 13 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in oligomenorrhea | 6 months
  The change in oligomenorrhea, i.e restoration of monthly menses or improvement in the menstrual pattern during 6 months while enrolled in the trial based on self report
Changes Vitamin D (25-hydroxyvitamin D) level | at enrollment, at 3 months after randomization and 6 months after randomization
  25-hydroxyvitamin D level will be measured by liquid chromatography-mass spectrometry (LC-MS/MS) or immunoassay

SECONDARY OUTCOMES:
Change in DHEAS level | at enrollment, at 3 months after randomization and 6 months after randomization
  The serum DHEA-S concentration is the traditional marker for adrenal androgen excession because it is produced almost exclusively by the adrenal glands and concentrations remain stable across the day and cycle. Preferred testing is done by immunoassay.
Changes in Androstenedione level | at enrollment, at 3 months after randomization and 6 months after randomization
  Androstenedione concentration assesses for hyperandrogenemia as well, it is produced by the ovary and the adrenal cortex and serves as precursor of testosterone. Data suggests that levels are elevated in approximately 20% of women with PCOS. Evaluation is done by Liquid Chromatography/Tandem Mass Spectrometry
Change in Anti-Mullerian hormone (AMH) level | at enrollment, at 3 months after randomization and 6 months after randomization
  AMH is a dimeric glycoprotein of the transforming growth factor-β superfamily that is involved in growth and differentiation of ovarian follicles. AMH is expressed in granulosa cells in the ovary and serves as a marker of ovarian reserve as well as marker of several ovarian pathologies such as PCOS, granulosa cell tumors and premature ovarian insufficiency. Level will be measured using Immunoassay (IA)
Change in testosterone level | at enrollment, at 3 months after randomization and 6 months after randomization
  Testosterone levels are elevated in vast majority of adolescents with PCOS. The free testosterone level is more sensitive for diagnosis of hyperandrogenic disorders compared with the total testosterone. Evaluation is done by Chromatography/Mass Spectrometry
Change in Hirsutism | at enrollment, at 3 months after randomization and 6 months after randomization
  Hirsutism is defined as excessive male-pattern facial and body hair. This will be measured by using the modified Ferriman Gallwey score by a provider with scores of less than 6 indicating no evidence of hirsutism, 6-8 indicating mild hirsutism, scores 8-15 indicating moderate hirsutism and scores greater than 15 indicating severe hirsutism.
Change Body Acne | at enrollment, at 3 months after randomization and 6 months after randomization
  European Dermatology Forum Guidelines group (2011) grading system will be used to describe acne in 4 areas of the body- face, upper chest, upper back, upper arms: minimal - comedonal acne, mild to moderate: moderate papulopustular acne, severe: severe papulopustular acne, moderate nodular acne; severe nodular acne,conglobate acne
Change in Facial | at enrollment, at 3 months after randomization and 6 months after randomization
  European Dermatology Forum Guidelines group (2011) grading system will be used to describe acne in 4 areas of the body- face, upper chest, upper back, upper arms: minimal - comedonal acne, mild to moderate: moderate papulopustular acne, severe: severe papulopustular acne, moderate nodular acne; severe nodular acne,conglobate acne

CONTACTS AND LOCATIONS:
Overall Officials: Alla Vash-Margita, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Children's Hospital, New Haven, Connecticut, United States